CLINICAL TRIAL: NCT06573203
Title: Clinical Effectiveness of Non-contact Heart Rate and Respiratory Rate Monitoring System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Jiaxing Yuanbeibei Technology Co. LTD (Unknown); Children's Hospital, Zhejiang University School of Medicine (Unknown)
Responsible Party: Principal Investigator, Shujun Li, Honorary Director of Nursing Department, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-IEC-0024-P-01
Record Dates: First submitted 2024-08-20; First posted 2024-08-27 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-08

CONDITIONS: Sleep; Infant，newborn; Vital Signs
Keywords: Sleep monitoring; Vital signs were monitored; Study of correlation
MeSH Terms: interventions — Respiratory Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Non-contact heart rate and respiratory rate monitoring system (Experimental): After admission, the non-contact mattress is placed under a normal mattress, and heart rate, respiratory rate, and sleep-related parameters can be collected through induction.
  Interventions: Device: Mindray ECG monitor; Device: aEEG; Other: Neonatal Sleep-Wake Assessment Tool (NSWAT) included four dimensions: eye movement, respiratory rate, facial expression and muscle activity.
- Electrocardiogram monitor (Active Comparator): Measuring vital signs
  Interventions: Device: Non-contact heart rate and respiratory rate monitoring system
- Amplitude-integrated EEG (Active Comparator): Sleep parameters were continuously measured by aEEG for 6 hours after admission.
  Interventions: Device: Non-contact heart rate and respiratory rate monitoring system
- Neonatal Sleep-Wake Assessment Tool (Active Comparator): It is suitable for all newborns to observe and evaluate the sleep phase, wake period and regularity, and guide the choice of care time. The scale includes four dimensions: eye movement, breathing rate, facial expression and muscle activity. The score range of each dimension is 0 ~ 2 points, and the score range is 0 ~ 8 points.
  Interventions: Device: Non-contact heart rate and respiratory rate monitoring system

INTERVENTIONS:
Device: Non-contact heart rate and respiratory rate monitoring system — Each neonate enrolled underwent four sleep and vital signs monitoring procedures after admission.
  Other Names: model YBB-B1
  Arms: Amplitude-integrated EEG; Electrocardiogram monitor; Neonatal Sleep-Wake Assessment Tool
Device: Mindray ECG monitor — Heart rate and respiratory rate of each enrolled child were monitored after admission.
  Other Names: model cPM 10C
  Arms: Non-contact heart rate and respiratory rate monitoring system
Device: aEEG — Each enrolled child underwent a 6-hour sleep-wake cycle, quiet sleep, and active sleep monitoring after admission.
  Other Names: model Nicolet EEG V32
  Arms: Non-contact heart rate and respiratory rate monitoring system
Other: Neonatal Sleep-Wake Assessment Tool (NSWAT) included four dimensions: eye movement, respiratory rate, facial expression and muscle activity. — The study nurses observed and scored the children's sleep-wake status 10 minutes after two meals during the mattress test period, each time for 5 minutes.
  Arms: Non-contact heart rate and respiratory rate monitoring system

SUMMARY:
In this study, hospitalized neonates were taken as the focus of the study. The non-contact heart rate and respiratory rate monitoring system was used to measure heart rate, respiratory rate, sleep parameters, ECG monitor, neonatal sleep-wake scale, amplitude-integrated electroencephalography. aEEG), in order to provide a theoretical basis for standardizing the operation of medical staff and formulating sleep protection strategies in the future, so as to promote the sleep quality of hospitalized neonates and improve the prognosis of neonates.

DETAILED DESCRIPTION:
The non-contact heart rate and respiratory rate monitoring system collected the body vibration signals of children through the heart rate and respiratory rate sensor, converted the pressure signals of vibration into electrical signals, extracted heart rate and respiratory rate, and extracted the characteristic parameters of sleep stages using heart rate and respiratory rate and body movement signals. It is characterized by no need to wear any equipment, the monitoring mattress is placed under the original baby mattress, no direct contact with the skin of the child, no comfort, and no change in the original sleep habits.

ELIGIBILITY:
Inclusion Criteria:

* Newborns admitted to our hospital for the first time, with gestational age ≥28w;
* Expected hospital stay ≥5 days.

Exclusion Criteria:

* Apgar score ≤3 at 1 or 5 min after birth;
* Severe congenital malformation; Severe hypoxic-ischemic encephalopathy, intraventricular hemorrhage of grade III and above; There were serious heart and lung diseases.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep-wake state | 10minutes after the meal, 5minutes each time, two times in total
  Sleep-wake state scores derived from a contact-free heart rate and respiratory rate monitoring system and NSWST measurements.
Number of sleep cycles | The hospital stay lasted 6 hours
  The number of sleep cycles obtained was monitored simultaneously by a non-contact heart rate and respiratory rate monitoring system and aEEG.
Proportion of quiet sleep | The hospital stay lasted 6 hours
  non-contact heart rate and respiratory rate monitoring system and aEEG were used to simultaneously measure the quiet sleep time for 6 hours, and then the proportion of quiet sleep was calculated.
Proportion of active sleep | The hospital stay lasted 6 hours
  non-contact heart rate and respiratory rate monitoring system and aEEG were used to simultaneously measure the active sleep time for 6 hours, and then the proportion of active sleep was calculated.

SECONDARY OUTCOMES:
Heart rate | The hospital stay lasted 6 hours
  Heart rate was measured simultaneously by non-contact heart rate and respiratory rate monitoring system and electrocardiogram monitor for 6 hours, and the average heart rate was calculated.
Respiratory rate | The hospital stay lasted 6 hours
  Respiratory rate was measured simultaneously by non-contact heart rate and respiratory rate monitoring system and electrocardiogram monitor for 6 hours, and the average respiratory rate was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhen Xu, Principal Investigator — The Children's Hospital Affiliated to the Medical College of Zhejiang University
Locations (1):
- The Children's Hospital Affiliated to the Medical College of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No